CLINICAL TRIAL: NCT06708832
Title: Pilot Study to Evaluate the Feasibility of Collecting Duodenal Fluid With SIMBA Capsules
Brief Title: To Evaluate the Feasibility of Collecting Duodenal Fluid With SIMBA Capsules
Acronym: CAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Nimble Science Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1266/2024
Record Dates: First submitted 2024-11-26; First posted 2024-11-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Liver Cirrhosis
Keywords: Microbiome; Metabolome; 16s rRNA; NMR; Pilot study; Duodenal microbiome; Liver Cirrhosis; SIMBA; Capsule; Metabolomics
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIMBA ingestion (Experimental): Participants will be prescreened for eligibility prior to obtaining informed consent. After informed consent is signed the participant will be screened and requested to complete a set of questionnaires prior to the ingestion of the SIMBA capsules. Then, a saliva and fecal sample will be collected and SIMBA capsules are ingested. The participant will be instructed on capsule ingestion. Retrieval of capsules occurs in their home environment. The participant is expected to continue searching their stool until both capsules are found. A fecal sample will be collected upon retrieval of first SIMBA capsule. After both capsules are collected the participants schedules an appointment to deliver the capsules to the study center and complete the second set of questionnaires. Additionally, saliva sample will be collected again.
  Interventions: Device: SIMBA ingestion

INTERVENTIONS:
Device: SIMBA ingestion — Ingestion of 2 SIMBA capsules at the same time and their excretion.
  Other Names: Small Intestine Microbiome Aspiration Capsules

SUMMARY:
In this study, the feasibility to use SIMBA (Small Intestinal MicroBiome Aspiration) capsules to collect small intestinal microbiome and metabolome information will be evaluated in patients with liver cirrhosis. Furthermore, the comparability oral, fecal and small intestinal microbiome and metabolome composition based on similarities and differences in 16s sequencing data and NMR metabolomics data will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Written informed consent
* Liver cirrhosis diagnosis by clinical/radiological/histological features
* Able to swallow a size-00 capsule (23mm length and 8mm width)

Exclusion Criteria:

* Inability to give informed consent
* Prior gastrointestinal disease, surgery, or radiation treatment which, in the Investigator's opinion, would lead to intestinal structuring or obstruction with a risk of capsule non-excretion, including, e.g., achalasia, eosinophilic esophagitis, cancer diagnosis or previous esophageal, gastric, small intestinal, or colonic surgery. Appendectomy or cholecystectomy more than 3 months before the screening visit is acceptable.
* History of known structural gastrointestinal abnormalities such as structures or fistulas leading to mechanical obstruction.
* Known history abdominal radiation treatment.
* Use of any medications in the week prior to the screening study visit, unless part of regular treatment, that could substantially alter gastrointestinal motor function (e.g., opioids, prokinetics, anticholinergics, GLP-1 analogues); laxative use is allowed if it is kept unchanged in the week prior to the study visit. Proton pump inhibitors (PPIs) are allowed provided a wash-out period of 48 h before swallowing SIMBA capsules and PPI treatment is resumed only 4 hours thereafter.
* Organic motility disorder, including gastroparesis, intestinal pseudo-obstruction, systemic sclerosis, Ogilvie's syndrome.
* Any significant heart, liver, lung, kidney, blood, endocrine or nervous system disease, which in the opinion of the investigator, would adversely affect study safety or outcome.
* History of oropharyngeal dysphagia, or other swallowing disorder with a risk of capsule aspiration.
* Antibiotic use (except for topical use) ≤ 12 weeks prior to screening. Potential participants may be eligible once a 12-week washout is completed.
* Consumption of probiotic or prebiotic supplements within 1 month prior to screening. Potential participants may be eligible once a 1-month washout is completed.
* Any prior Fecal Microbiota Transplantation.
* Colon cleanses/bowel prep for 2 weeks
* Pregnant or breastfeeding.
* Planning to become pregnant.
* Are scheduled for an MRI at any time during the study. Potential participants may be eligible to participate once their MRI procedure is completed.
* History of less than three (3) bowel movements per week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of capsules successfully recovered | From ingestion of capsules to their excretion
  Number of capsules successfully recovered with sufficient amount of fluid collected for the analysis (absolute number, percentage)

SECONDARY OUTCOMES:
Composition of the microbiome in capsule fluid (16s rRNA) | From ingestion of capsules to their excretion
  Composition of the microbiome in capsule fluid measured by 16s rRNA sequencing
Composition of the microbiome in stool (16s rRNA) | From ingestion of capsules to their excretion
  Composition of the microbiome in stool microbiome measured by 16s rRNA sequencing
Composition of the microbiome in saliva (16s rRNA) | From ingestion of capsules to their excretion
  Composition of the microbiome in saliva microbiome measured by 16s rRNA sequencing
Composition of the metabolome in capsule fluid (NMR) | From ingestion of capsules to their excretion
  Composition of the metabolome in capsule fluid measured by NMR metabolomics
Composition of the metabolome in saliva (NMR) | From ingestion of capsules to their excretion
  Composition of the metabolome in saliva measured by NMR metabolomics
Composition of the metabolome in stool (NMR) | From ingestion of capsules to their excretion
  Composition of the metabolome in stool measured by NMR metabolomics
Number of adverse events | From ingestion of capsules to their excretion

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer-Köllner, Assoc. Prof., Principal Investigator — Medical University of Graz Department of Gastroenterology and Hepatology Auenbruggerplatz 15 8036 Graz
Locations (1):
- Department of Internal Medicine, Division of Gastroenterology and Hepatology, Liver study clinic, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided